CLINICAL TRIAL: NCT03985644
Title: Multi-center Clinical Application of Hangzhou Criteria in Liver Transplant Candidate Selection for Hepatocellular Carcinoma
Brief Title: Multi-center Clinical Application of Hangzhou Criteria in Liver Transplantation for Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, professor, Zhejiang University
Other Study IDs: zju2017xux
Record Dates: First submitted 2019-06-10; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: HCC; Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fulfilling Hangzhou criteria: Patients flfilling Hangzhou critieria:
  Without macrovascular invasion Tumor burden <=8 cm Preoperative AFP level <=400 ng/mL Histopathologic grades I, II
- Exceeding Hangzhou criteria: Patients exceeding Hangzhou critieria

SUMMARY:
Liver transplantation is an optimal radical therapy for selected patients with hepatocellular carcinoma. Hangzhou criteria could safely and effectively expand Milan criteria with expanded population and comparable survival. The purpose of this study was to evaluate the Hangzhou criteria in a multi-center cohort.

DETAILED DESCRIPTION:
Liver cancer is the sixth most commonly diagnosed cancer and the fourth leading cause of cancer-related deaths worldwide. Among all the liver cancer cases, hepatocellular carcinoma (HCC) constitutes 75-85%. Liver transplantation is the most effective treatment for HCC and is in high demand in China. The advent of Milan criteria has helped to select the recipients reasonably. However, the organ allocation system driven by the Milan criteria seemed to be too strict so that many centers worldwide have expanded the criteria in the aspects of morphological features, histopathology and biomarkers. Hangzhou criteria introduce the covariables of histopathologic grading and α-fetoprotein (AFP) into the selection of recipients for the first time. Based on the multi-center HCC patient cohort undergoing transplantation, this study aims to characterize an ideal candidate selecting system beyond the Milan criteria.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years and <=75 with HCC confirmed by histopathology;
* Undergoing a primary whole or split liver transplant from a deceased donor;

Exclusion Criteria:

* Incomplete follow-up;
* Missing essential data for analysis (tumor size, number, differentiation grade, α-fetoprotein (AFP)) ;
* Vascular invasion according to radiological criteria;
* Perioperative mortality (<30 days) ;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years and <=75 with HCC who underwent a primary whole or split liver transplant from a deceased donor were eligible for enrollment at the time of transplant. All of patients were histologically confirmed HCC by postoperative pathological examination in the participating centers. The donor-to-recipient arrangements all conformed to the principle of ABO compatibility. Key exclusion criteria were incomplete follow-up, missing essential data for analysis (tumor size, number, differentiation grade, α-fetoprotein (AFP)) or vascular invasion according to radiological criteria, and excludes those with perioperative mortality (<30 days)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival

SECONDARY OUTCOMES:
Recurrence rate | 5 years
  Recurrence rate